CLINICAL TRIAL: NCT01866254
Title: Use of Intrathecal Hydromorphone in Elective Cesarean Deliveries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grace Shih, MD (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor-Investigator, Grace Shih, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13527
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: Hydromorphone; Morphine; cesarean delivery; pain management; respiratory depression
MeSH Terms: conditions — Pain; Agnosia; Respiratory Insufficiency | interventions — Hydromorphone; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydromorphone (Experimental): 100 mg, intrathecal administration
  Interventions: Drug: Hydromorphone
- Morphine (Active Comparator): 200 mg, intrathecal administration
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Hydromorphone — Injection of 100 mcg hydromorphone into the intrathecal space
  Other Names: DILAUDID® INJECTION
  Arms: Hydromorphone
Drug: Morphine — Injection of 200 mcg of intrathecal morphine
  Other Names: Duramorph
  Arms: Morphine

SUMMARY:
The purpose of this study is to determine if intrathecal hydromorphone will relieve pain as well as intrathecal morphine after cesarean delivery, with fewer side effects.

DETAILED DESCRIPTION:
Intrathecal morphine has long been the standard pain medication used in cesarean sections. Since some patients cannot tolerate morphine, hydromorphone may be an acceptable alternative. Intrathecal Intrathecal hydromorphone has been shown to be effective at treating post cesarean section pain and possibly with less side effects than morphine.

One side effect of morphine is respiratory depression occurring hours after the start of morphine use. Respiratory depression occurs when air being taken into the lungs is less than normal, leading to a lower amount of oxygen and carbon dioxide being exchanged in the blood stream. Because hydromorphone dosages are lower and it has a quicker onset of action than morphine, it is believed that the use of hydromorphone should decrease the possibility of delayed respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective Cesarean sections under spinal anesthesia or combined spinal anesthesia
* ASA status of I-III
* BMI < 40
* Able to understand and sign informed consent

Exclusion Criteria:

* Severe pre-eclampsia
* Conversion to general anesthetic
* History of chronic opioid use
* Allergy to morphine, or hydromorphone
* Hyperemesis gravidarum
* Emergency case
* Patients who have an infection at the intended site of spinal insertion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12-04 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores | from Baseline to 24 Hours
  Pain scores to be measured using the verbal response scale (VRS). The VRS pain score is measured on a scale of 0-10 with 0 representing absolutely no pain and 10 representing worst pain imaginable

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to 24 Hours
  Patients will be monitored hourly for first 12 hours followed by every 2 hours for the next 12 hours. Masimo acoustic monitor will monitor respirations.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Shih, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States